CLINICAL TRIAL: NCT06920160
Title: Determination of the Efficacy of Remote Monitoring of Patients With Heart Failure and Reduced Ejection Fraction Using Caaring® Software
Brief Title: Efficacy of Remote Monitoring of Patients With Heart Failure and Reduced Ejection Fraction by Using Caaring® Software
Acronym: (CAARdioRING)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Persei Vivarium (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAARdioRING
Record Dates: First submitted 2025-03-25; First posted 2025-04-09 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure; Reduced Ejection Fraction; DTx; Caaring; remote patients monitoring; Digital Health
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online telemonitoring group (G_CAARING) (Active Comparator): The monitoring and control of these patients will be carried out remotely through the Caaring® platform. Patients will connect to an APP on a mobile phone. They will have to complete the data and questionnaires related to the study variables.
  Interventions: Device: software Caaring (remote monitoring app)
- Control Group (G_Control) (No Intervention): The data of these patients are collected prospectively from their routine medical visits for 12 weeks after inclusion

INTERVENTIONS:
Device: software Caaring (remote monitoring app) — Caaring is an electronic data collection notebook that allows patients to confidentially fill out data/ questionnaires on their mobile phone and report them through an application that will be installed on the patient's mobile phone. Besides, This group (G_CAARING) will receive educational and prevention recommendations relative to Heart Faillure.
  Arms: Online telemonitoring group (G_CAARING)

SUMMARY:
The goal of this clinical trial investigation with device is to determinate the effectiveness of remote monitoring of patients with heart failure with reduced ejection fraction heart (EFS40%) using Caaring® software.

The main question it aims to answer is if the development of a self-management platform (Caaring®) that enhances the role of the patient with heart failure in the course of their disease will reduce the number of re-entries. For this, researchers will compare the assessments between the two groups.

This is a randomized study with two arms. Online telemonitoring group: The follow-up of these patients will be carried out prospectively remotely through the Caaring® platform. And Prospective Control group: The data of these patients are collected prospectively for their routine medical visits for 12 weeks after their inclusion.

In addition, Control group patients must have clinical data from the 12 weeks after to their inclusion date available in the Medical Record, and/or through the monitoring platforms of the continuous monitoring devices.

Participants with heart failure will continue to receive conventional care and must have sufficient technological skills to use a smartphone.

DETAILED DESCRIPTION:
This is a longitudinal, comparative non-inferiority, multicenter, with 2 arms Medical Device Clinical Trial.

The protocol and informed consent documents have been reviewed and approved by the hospital human subjects reviewboard and the study will be performed in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients diagnosed with heart failure with reduced ejection fraction (EFS40%)
* Patients discharged after an episode of acute heart failure and/or patients who are being followed up after being admitted for heart failure.
* Patients who extensively use a smartphone.
* lnformed Consent is obtained from the patient

Exclusion Criteria:

* Patients with cognitive ar sensory difficulties or with insufficient command of Spanish who, in the opinion of the investigator, makes it difficult to understand the questions ar the scales, as long as they do not have a legally authorized representative capable of participating in the study.
* Transient patients in whom it may be anticipated that follow-up will not be completed due to a change of residence.
* Patients Who are participating at the time of recruitment in any other clinical trial. Participation in observational studies will not be an exclusion criteria.
* Patients whose main diagnosis is a poorly controlled mental disorders ar other medical illness.
* Patients with terminal illness and/or in palliative care according to the criteria of the SECPAL (Spanish Society of Palliative Care).
* lnstitutionalized patients
* Patients who are pregnant ar breastfeeding.
* Patients whose inclusion is not considered advisable by the investigator's assessment due to they are under specific follow-up in other hospital units (hemodialysis, transplants, etc.) that require mandatory hospital attendance less frequently than once every two months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of re-entries in patients with heart failure | Day 0, Week 12
  Number of re-entries in patients with heart failure

SECONDARY OUTCOMES:
Changes in Health-related quality of life (WHOQOL) | Day 0, Week 12
  Change in the patient's quality of life scale the study comparad to baseline: WHOQOL questionnaire (Value 0- 100). A higher score reflects a higher health-related quality of life.
Adherence treatment equal to or greater than 80% | Day 0 and Weekly up to 12 weeks
  Percentage of patients with treatment adherence for heart failure equal to or greater than 80%
Changas in the patient's MEDAS scale: Adherence to Mediterranean Diet | Day 0, Week 12
  Changes in patient's scale MEDAS (Mediterranean Diet Adherence Screener) scores at week 4 and at the end of the study compared to baseline. Values: 0-14, a higher score reflects a better adherence to the Mediterranean Diet.
Changes in the patient's Clinical Data | Day O, every 3 days up to Week 12
  Changes in patient's Clinical data (symptoms related to heart failure) measured through a specific form created for this purpose.
Patient satisfaction with the software Caaring | Week 12
  The patient satisfaction will be measured through a specific satisfaction questionnaire created for this purpose. (Value 3-15). A higher score reflects greater satisfaction with software care.
Changes in the patient's in Liquid Consumption | Day 0, Week 12
  Changes in patient's Liquid Consumption Questionnaire. The changes will be measured through a specific form created for this purpose
Adherence treatment equal to 100% | Day 0 and Weekly up to 12 weeks
  Percentage of patients with treatment for heart failure adherence equal to 100%

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, A Coruña
  - Hospital Universitario de Son Llatzer, Palma de Mallorca, Balearic Islands

IPD SHARING:
Plan to Share IPD: No